CLINICAL TRIAL: NCT06871930
Title: Characteristic and Survival Outcomes in Hepatocellular Carcinoma Patients: on Top of Viral Hepatitis Versus Combined Viral and Metabolic-Associated Steatotic Liver Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mamdouh Ali kamel Ibrahim Badary, residant doctor, Assiut University
Other Study IDs: HCC viral Vs MASLD hepatitis
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: HCC patients with viral hepatitis alone (HBV or HCV).
- Group 2: HCC patients with combined viral hepatitis (HBV or HCV) and MASLD.

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most prevalent cancers globally and ranks as the third leading cause of cancer-related deaths . It primarily arises in patients with chronic liver disease and liver cirrhosis, which can result from various etiologies, including viral hepatitis and metabolic disorders. Viral hepatitis, especially Hepatitis B virus (HBV) and Hepatitis C virus (HCV), is well-established as a major risk factor for HCC. Chronic HBV infection is associated with a higher risk of HCC, particularly in areas with high endemicity . Similarly, HCV is linked to significant liver-related morbidity and mortality, with HCC being a leading complication .

In recent years, the increasing prevalence of metabolic-associated steatotic liver disease (MASLD) has emerged as a significant contributor to liver disease and HCC, particularly in the context of the obesity epidemic. MASLD is characterized by fatty liver disease associated with metabolic risk factors such as obesity, insulin resistance, and type 2 diabetes . The combination of chronic viral hepatitis and MASLD may exacerbate liver damage and contribute to the development of HCC, although the specific mechanisms remain to be fully elucidated Despite the known associations between these risk factors and HCC, there remains a shortage of comprehensive studies comparing the clinical characteristics and survival outcomes of patients with HCC due to viral hepatitis alone versus those with combined viral and MASLD. Understanding these differences is crucial for optimizing surveillance, treatment strategies, and prognostic assessment for patients at risk of HCC.

the aim of the study Compare the clinical characteristics of HCC patients with viral hepatitis versus those with combined viral and MASLD.

- Analyze survival outcomes in both groups and correlate these outcomes with patients' characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) diagnosed with HCC based on radiological, histological (if needed), or biomarker criteria (e.g., elevated AFP).

  . Documented history of:
* Chronic Hepatitis B virus (HBV) infection or Hepatitis C virus (HCV) infection.
* MASLD defined as hepatic steatosis (≥5%) confirmed by FibroScan or abdominal ultrasound along with at least one metabolic risk factor (e.g., obesity, type 2 diabetes, hypertension).

Ability to provide informed consent

Exclusion Criteria:

* . Other causes of chronic liver disease (e.g., autoimmune hepatitis, hemochromatosis, Wilson's disease).
* Patients with incomplete clinical or diagnostic data.
* Presence of other malignancies.
* Patients refuse to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HCC patients divided into two group:
  * Group 1: HCC patients with viral hepatitis alone (HBV or HCV).
  * Group 2: HCC patients with combined viral hepatitis (HBV or HCV) and MASLD.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 1 year
  Comparison of overall survival between HCC patients with viral hepatitis alone and those with combined viral hepatitis and MASLD, measured from diagnosis to death or last follow-up.